CLINICAL TRIAL: NCT00535028
Title: A Phase IIa Study To Investigate The Effects of AER 001 on Antigen Challenge In Atopic Asthmatic Subjects Following Repeated Administration.
Brief Title: A Phase IIa Study of Subcutaneous AER 001 on Antigen Challenge In Atopic Asthmatic Subjects (28 Day Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerovance, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QGUY/2004/IL4-13/-01; EUDRACT 2004-002836-25
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Allergic Asthma
Keywords: asthma; allergy; interleukin-4; interleukin-13; IL-4; IL-13; atopic; late asthmatic response; inflammation
MeSH Terms: conditions — Asthma; Hypersensitivity; Rhinitis, Allergic; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AER 001 s.c. once daily for 28 days
  Interventions: Drug: AER 001
- P (Placebo Comparator): placebo s.c. once daily for 28 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AER 001 — AER 001 25 mgs s.c. once daily for 28 days
  Arms: A
Drug: placebo — sterile saline
  Arms: P

SUMMARY:
This is a single center, double-blind, randomised parallel group design study to investigate the effects of AER 001 on the late phase asthmatic resonse in asthmatic subjects. AER 001 is to be administered subcutaneously (25 mg, once daily) for 28 days. The asthmatic subjects will be challenged with allergen both before and after AER 001 treatment (at screen and at Day 28). The primary outcome will be late phase sthmatic response (the max drop in FEV1 from 4-10 hours after an allergen challenge).

DETAILED DESCRIPTION:
Objectives:

Primary Objective

* To investigate the late asthmatic response in mild to moderate asthmatics.. Secondary Objectives
* To examine the effects of AER 001 on cutaneous antigen response, antigen induced airway hyperactivity and sputum eosinophilia.

Methodology: Study Design:

* Single centre, phase IIa, double-blind, randomised, parallel group, repeated dose study in male and female asthmatic subjects.
* A sufficient number of subjects (at least 24 subjects) will be recruited to ensure that at least 20 completed sets of data will be obtained.
* Subjects will be randomised to receive either AER 001 25 mg / Placebo in a ratio of 1 active : 1 placebo.
* Treatments will be administered as a sub-cutaneous injection.
* Subjects are to receive a daily administration of AER 001 / placebo over a 4 week period.
* Subjects will be admitted to the unit at least 2 hours prior to the first dose administration. On the first dosing occasion the subjects will remain in the unit under clinical supervision for at least 30 minutes post dose or until the Investigator is satisfied for them to be discharged. On subsequent dosing days the subjects will be admitted to the unit at least 45 minutes prior to dosing and remain in the unit for at least 15 minutes post dose or until the Investigator is satisfied for them to be discharged.

ELIGIBILITY:
Inclusion Criteria:

* • Adult males and females > 18 years.

  * Subjects who if female, are not currently pregnant or breast feeding and are using medically acceptable methods of contraception.
  * Subjects who have a pre study medical history, physical examination, 12 Lead ECG acceptable to the investigator.
  * Subjects who have clinical laboratory tests within the reference ranges or clinically acceptable to the investigator.
  * Subjects who are negative for HbsAg, hepatitis C antibody and HIV II and I test at screening.
  * Subjects who are negative for drugs of abuse and alcohol tests at screening and admission.
  * Positive response on screening to a skin prick test.
  * Subjects who respond < 8 mg / mL on the methacholine challenge.
  * Subjects, who on the Allergen challenge, have a PC20 on allergen and exhibit a late phase response (>or = 15% between 4-10h) following the allergen challenge.
  * Subjects who have a FEV1 >70% of predicted.
  * Have not received steroid treatment in the prior month.
  * Subjects who are non-smokers for at least 3 months prior to screening.
  * Have a < 10 pack year history.
  * Satisfies the Global Initiative in Asthma (GINA, 2002) definition of asthma or have been on treatment for asthma.
  * Subjects with stable, adequately treated medical conditions may be enrolled provided the Principal Investigator does not consider their study participation to place them at increased risk of adverse events. Subjects should continue their concomitant treatments without change during the study.
  * Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

* • Subjects who do not conform to the above inclusion criteria.

  * Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders. Which would preclude antigen challenge
  * Subjects who have a clinically relevant surgical history. Which would preclude antigen challenge
  * Subjects who have a clinically relevant family history. Which would preclude antigen challenge
  * Subjects who have a history of relevant drug hypersensitivity.
  * Subjects who have a history of alcoholism.
  * Subjects who have a history of drug abuse.
  * Subjects who consume more than 28 units of alcohol a week. (unit = 1 glass of wine = 1 measure of spirits = ½ pint of beer)
  * Subjects who have a significant infection or known inflammatory process on screening.
  * Subjects who have acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn)
  * Subjects who have an acute infection such as influenza at the time of screening and/or admission.
  * Female subjects who are not using an acceptable method of contraception.
  * Subjects who have used any investigational drug and /or participated in any clinical trial within 3 months of their first dosing.
  * Subjects using medication, which in the opinion of the Investigator will affect the outcome of the study.
  * Subjects who have donated and/or received any blood or blood products within the previous 3 months prior to first dosing (to review on a case by case basis).
  * Subjects who cannot communicate reliably with the investigator.
  * Subjects who are unlikely to co-operate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Max %fall in FEV1 during the late phase asthmatic response (4-10 hours after allergen challenge) | After 28 days of treatment with study medication

SECONDARY OUTCOMES:
To examine the effects of AER 001 on cutaneous antigen response, antigen induced airway hyperactivity and sputum eosinophilia. | After 28 days of treatment with study medication

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, M.D., Principal Investigator — Guy's Drug Research Unit, Quintiles, Ltd.
Locations (1):
- Guy's Drug Research Unit, Quintiles, Ltd., 6 Newcomen Street London, London, United Kingdom

REFERENCES:
- [Derived] Wenzel S, Wilbraham D, Fuller R, Getz EB, Longphre M. Effect of an interleukin-4 variant on late phase asthmatic response to allergen challenge in asthmatic patients: results of two phase 2a studies. Lancet. 2007 Oct 20;370(9596):1422-31. doi: 10.1016/S0140-6736(07)61600-6. PMID 17950857